CLINICAL TRIAL: NCT02670512
Title: Assessment of Telehome Monitoring in Patients on Peritoneal Dialysis (CONNECT Trial): A Multicentre Randomized Controlled Trial
Brief Title: Assessment of Telehome Monitoring in Patients on Peritoneal Dialysis: A Multicentre Randomized Controlled Trial
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Connect1.13
Record Dates: First submitted 2016-01-18; First posted 2016-02-01 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2020-11

CONDITIONS: End-Stage Renal Disease
Keywords: End-Stage Renal Disease; Peritoneal Dialysis; Telehomecare; Telehome Monitoring
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehome Monitoring (Experimental): Patients in this arm will use the telehome monitoring device (a mobile tablet) to support them with their peritoneal dialysis (communication, treatment tracking, supply tracking, appointment reminders, educational content).
  Interventions: Device: Telehome Monitoring
- Standard of Care (No Intervention): Patients in this arm use the standard of care for peritoneal dialysis, which is simple telephone communication and using pen and paper log to track their treatments and supplies.

INTERVENTIONS:
Device: Telehome Monitoring
  Other Names: eQ Connect™
  Arms: Telehome Monitoring

SUMMARY:
Compared to hemodialysis, patients on peritoneal dialysis live longer and healthier, have a higher quality of life and cost approximately $40,000 less to the healthcare system per patient per year. However, only 18% of dialysis patients in Canada currently use peritoneal dialysis because patients often feel isolated from the healthcare team and lack the confidence to manage treatments by themselves. This study will assess a telehome monitoring system (eQ Connect™), allowing for up-to-date data transmission and digital interaction between the patients at home and their healthcare team. From the patients' perspective, this technology is an easier way to communicate with their healthcare providers, track their treatment and supplies, and receive training and support. From the providers' perspective, eQ Connect™ delivers up-to-date patient data and provides an efficient way to keep track of the patients' progress. This intervention has the potential to improve the patients' clinical outcomes, quality of life, reduce the costs of dialysis to the healthcare system and ultimately empower patients to start and stay on peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent
2. Patient or primary care giver able to read and speak English
3. Over 18 years of age
4. Patient on PD (APD/CAPD) for at least 3 months
5. Patient or primary care giver cognitively and physically capable and willing to interact with a tablet computer and perform self-measurements (e.g. taking weight)

Exclusion Criteria:

1. Scheduled kidney transplant within 1 year (identified, processed and medically worked out their donor)
2. Life expectancy <1 year (estimated by physician)
3. In long-term care facility
4. Deemed unable to comply with the telehome monitoring support system (e.g. due to vision problems, literacy, lack of manual dexterity to accurately interact with the tablet, or decreased cognitive function such as memory loss) by physician
5. Participating in another interventional trial that could influence the intervention or outcome of this trial
6. Was in another interventional trial that could influence the intervention or outcome of this trial, ≤4 weeks prior to recruitment
7. Patients on hybrid dialysis (those on both peritoneal dialysis and hemodialysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Composite clinical outcome | 1 year (plus 12 weeks for complete follow-up of technique failure)
  The primary outcome is a composite of technique failure (switching to hemodialysis for ≥12 weeks), infections (peritonitis, exit-site, tunnel) and hospital encounters (ER visits, hospitalizations).

SECONDARY OUTCOMES:
Health-related Quality of Life | 1 year
  This study will utilize the Kidney Disease Quality of Life-36 (KDQOL-36) Instrument and EQ-5D to assess HRQOL.
Time spent communicating | 1 year
  This measure captures the time a patient spends communicating with the healthcare team. This is measured through automated telephone logs and paper telephone logs that are documented by nurses. For patients in the intervention arm, investigators will also obtain the duration of video calls and amount of time spent on the message screen (number of minutes). We will also capture the number of messages that are sent on the telehome monitoring device.
Number of missed appointments | 1 year
  Investigators will examine the number of appointments that a patient has missed, which is documented through a scheduling software from the clinic.
Nurse Overtime hours | 1 year
  Investigators deliver care for the patients. The number of hours worked over-time are documented in a telephone log manually, which includes the patient's name, reason for call and call duration.
Number of clinic visits | 1 year
  The number of clinic visits will be collected through scheduling software from the PD clinic.
Hospitalization Days | 1 year
  Investigators will compare the length of hospitalizations (in days) between intervention and control group.
Nursing Costs | 1 year
  Investigators will compare costs by applying each centre's hourly nursing cost to the number of hours nurses spent communicating with the patient (derived from "time spent communicating" measure).
Healthcare Utilization Costs | 1 year
  Investigators will use the Case Costing Macro at ICES to compare the health utilization costs between two groups, including costs from emergency room visits and hospitalizations. (This is only applicable to the Ontario Centres).
Dialysis Supplies Costs | 1 year
  Investigators will compare the cost of supplies between the intervention and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Arsh K Jain, MD, Principal Investigator — University of Western Ontario, Canada
Locations (11):
- Canada (11):
  - Royal Columbian Hospital - Fraser Health Authority, New Westminster, British Columbia
  - Seven Oaks General Hospital, Winnipeg, Manitoba
  - QEII Health Sciences Centre - Nova Scotia Health Authority, Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Trillium Health Partners - Mississauga Hospital, Mississauga, Ontario
  - Mackenzie Health, Richmond Hill, Ontario
  - Scarborough Health Network - General Hospital, Scarborough Village, Ontario
  - Humber River Hospital, Toronto, Ontario
  - St. Paul's Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Jeffs L, Jain AK, Man RH, Onabajo N, Desveaux L, Shaw J, Hensel J, Agarwal P, Saragosa M, Jamieson T, Wong I, Maione M, Bhatia RS. Exploring the utility and scalability of a telehomecare intervention for patients with chronic kidney disease undergoing peritoneal dialysis-a study protocol. BMC Nephrol. 2017 May 10;18(1):155. doi: 10.1186/s12882-017-0557-y. PMID 28486991